CLINICAL TRIAL: NCT03785184
Title: A Phase 2, Multicenter, Single Arm, Open Label Study of Venetoclax Plus Lenalidomide and Dexamethasone for the Treatment of Newly Diagnosed t(11;14)-Positive Multiple Myeloma in Subjects Who Are Ineligible for High-Dose Therapy
Brief Title: A Study of Venetoclax Plus Lenalidomide and Dexamethasone for the Treatment of Newly Diagnosed t(11;14)-Positive Multiple Myeloma in Subjects Who Are Ineligible for High-Dose Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-104
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cancer; t(11;14)-Positive Multiple Myeloma; Venetoclax; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — venetoclax; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Lenalidomide + Dexamethasone (Experimental): Venetoclax up to 800 mg orally every day (QD) QD on Days 1 - 28 plus lenalidomide up to 25 mg orally QD on Days 1 - 21 (28 day cycle) plus dexamethasone up to 40 mg orally once weekly (QW).
  Interventions: Drug: venetoclax; Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: venetoclax — tablet; oral
  Other Names: ABT-199
Drug: lenalidomide — capsule; oral
  Other Names: Revlimid
Drug: dexamethasone — tablet; oral

SUMMARY:
This study will evaluate the safety and preliminary efficacy of venetoclax when combined with lenalidomide and dexamethasone for participants with newly diagnosed, active t(11;14) positive multiple myeloma (MM).

This study will consist of 2 parts: Part 1 Dose Escalation and Part 2 Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

* Must have documented, confirmed active multiple myeloma (MM) with greater than or equal to 10% clonal bone marrow plasma cells or biopsy-proven bone or extramedullary plasmacytoma and any one or more of the following myeloma-defining events:

  * Evidence of end organ damage attributed to the underlying plasma cell proliferative disorder and satisfying at least one of the protocol specified laboratory criteria for calcium elevation, renal failure, anemia, or lytic bone lesions; OR
  * One or more of the biomarkers of malignancy as described in the protocol.
* Must have MM positive for the t(11;14) translocation, as determined by methods described in the protocol.
* Must have measurable disease defined by at least one of the following criteria:

  * Serum M-protein ≥ 1.0 g/dL (immunoglobulin [Ig]G myeloma) or greater than or equal to 0.5 g/dL (IgA, IgM, IgD, or IgE myeloma);
  * Urine M-protein greater than or equal to 200 mg/24 hours;
  * Serum free light chain (FLC) greater than or equal to 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal.
* Newly diagnosed and not considered a candidate for high-dose therapy and hematopoietic stem cell transplantation (HSCT)
* Must have Eastern Cooperative Oncology Group performance status less than or equal to 2.

Exclusion Criteria:

* Has a co-existing condition as specified in the protocol.
* Has history of other active malignancies, including myelodysplastic syndromes (MDS) within the past 3 years with specific exceptions detailed in the protocol.
* Has been treated with or received any of the following:

  * Prior or current systemic therapy or hematopoietic stem cell transplantation (HSCT) for MM (a short course of treatment with corticosteroids equivalent to dexamethasone 40 mg/day for a maximum of 4 days is allowed before treatment); use of systemic strong or moderate inhibitor or inducer of cytochrome P450(CYP)3A within 7 days before the first dose of study drug.
  * Radiation therapy within 2 weeks of dosing
  * Plasmapheresis within 4 weeks of dosing
  * Immunization with live vaccine within 8 weeks of dosing
* Has a contraindication or inability to comply with antithrombotic prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-29 (Estimated); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participates Who Achieve CR | From baseline up to approximately 24 months
  Complete response (CR) is defined as negative immunofixation of serum and urine, and disappearance of any soft tissue plasmacytomas, and < 5% plasma cells in bone marrow.

SECONDARY OUTCOMES:
Percent of Participants Who Achieve MRD Negativity | From baseline up to approximately 24 months
  Minimal residual disease (MRD) negative after treatment is described as less than one myeloma cell per 100,000 bone marrow cells.
Percent of Participants Who Achieve VGPR or Better | From baseline up to approximately 24 months
  Very Good Partial Response (VGPR) per international myeloma working group (IMWG) criteria is defined as serum or urine myeloma protein (m-protein) detectable by immunofixation but not on electrophoresis, or greater than or equal to 90% reduction in serum m-protein and urine m-protein less than 100 mg/24 hours.
Overall Response Rate (ORR) | From baseline up to approximately 24 months
  ORR is described as the percentage of participants who experience partial response (PR) or better; PR per IMWG is described as follows:
  * ≥ 50% reduction of serum M-protein and reduction in 24-hour urinary M protein by ≥ 90% or to < 200 mg/24 h
  * If the serum and urine M-protein are not measurable, a decrease ≥ 50% in the difference between involved and uninvolved free light chain (FLC) levels is required in place of the M-protein criteria
  * If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, ≥ 50% reduction in bone marrow plasma cells is required in place of M-protein, provided baseline percentage was ≥ 30%
  * In addition, if present at baseline, ≥ 50% reduction in size of soft tissue plasmacytomas is also required
Time to Response (TTR) | From baseline up to approximately 24 months
  Time to response is defined as the time from randomization to the first response (CR, stringent complete response [sCR], VGPR, PR).
Duration of response (DOR) | Approximately 7 years
  DOR is defined as the time from first observation of PR to the time of disease progression, with deaths from causes other than progression censored.
Progression-free Survival (PFS) | Approximately 7 years
  PFS is defined as time from start of the treatment to disease progression or death (regardless of cause of death), whichever comes first.
Minimal Residual Disease (MRD) Negativity Rate at 12 Months | Approximately 12 months after initial dose of study drug
  Percent of participants meeting the MRD Negative criteria at 12 months after initial dose; MRD Negative defined as less than one myeloma cell per 100,000 bone marrow cells.
Time to Disease Progression (TTP) | Approximately 7 years
  TTP is defined as the time from start of treatment to disease progression, with deaths from causes other than progression censored.
Time to Next Treatment (TTNT) | Approximately 7 years
  The time to next treatment is defined as the time between the date of the first study drug intake and the date of the first next treatment intake after study drug discontinuation.
Overall Survival (OS) Rate | Approximately 7 years
  OS was defined as the time from the date the participant was randomized to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (22):
- United States (7):
  - City of Hope /ID# 212211, Duarte, California
  - Marin Cancer Care /ID# 208476, Greenbrae, California
  - University of California, Los Angeles /ID# 208516, Los Angeles, California
  - Karmanos Cancer Institute /ID# 208805, Detroit, Michigan
  - Henry Ford Hospital /ID# 208481, Detroit, Michigan
  - Duke University Hospital /ID# 208306, Durham, North Carolina
  - UPMC Hillman Cancer Ctr /ID# 208121, Pittsburgh, Pennsylvania
- Australia (5):
  - Westmead Hospital /ID# 210267, Westmead, New South Wales
  - Flinders Centre for Innovation /ID# 210697, Bedford Park, South Australia
  - St. Vincents Hosp Melbourne /ID# 210266, Fitzroy, Victoria
  - Austin Hospital /ID# 210268, Heidelberg, Victoria
  - Monash Medical Centre /ID# 210269, Melbourne, Victoria
- Canada (4):
  - Tom Baker Cancer Centre /ID# 208549, Calgary, Alberta
  - Princess Margaret Cancer Centr /ID# 208923, Toronto, Ontario
  - Hopital Maisonneuver-Rosemont /ID# 208550, Montreal, Quebec
  - McGill Univ HC /ID# 208486, Montreal, Quebec
- Spain (6):
  - Clinica Universitar de Navarra - Pamplona /ID# 209883, Pamplona, Navarra, Comunidad
  - Hospital Clinic de Barcelona /ID# 209888, Barcelona
  - Hspital Universitario Gregorio Maranon /ID# 209926, Madrid
  - Clinica Universitar de Navarra - Madrid /ID# 210131, Madrid
  - Hosp Univ 12 de Octubre /ID# 209887, Madrid
  - Hospital Univ Dr. Peset /ID# 209884, Valencia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://www.rxabbvie.com